CLINICAL TRIAL: NCT01784926
Title: Late Dislocation of Intraocular Lens (IOL) Following Cataract Surgery: an Evaluation of Two Different Surgical Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marius Dalby, MSc, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1981
Record Dates: First submitted 2013-01-29; First posted 2013-02-06 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Intraocular Lens Dislocation
Keywords: cataract surgery; scleral suturing; Verisyse; Late in-the-bag IOL dislocation

STUDY DESIGN:
Masking Description: Investigator masked for group affiliation during image analysis
Oversight: Data Monitoring Committee: No

ARMS (2):
- IOL repositioning (Other): Operation method: Intraocular lens repositioning by scleral suturing
  Interventions: Procedure: Intraocular lens repositioning by scleral suturing
- IOL exchange (Other): Operation method: Intraocular lens exchange with retropupillary iris-claw lens
  Interventions: Procedure: Intraocular lens exchange with retropupillary iris-claw lens

INTERVENTIONS:
Procedure: Intraocular lens repositioning by scleral suturing
  Arms: IOL repositioning
Procedure: Intraocular lens exchange with retropupillary iris-claw lens
  Arms: IOL exchange

SUMMARY:
A prospective randomized study on patients with late in the bag intraocular lens (IOL) dislocation, after cataract surgery. To obtain normal visual function, these patients needs surgery. In this study the investigators will look for advantages and dis-advantages after two different surgical approaches to late in-the-bag IOL dislocation.

DETAILED DESCRIPTION:
In this prospective, randomized study The investigators will include at least 80 patients with late intraocular lens (IOL) dislocation in the capsular complex, after cataract surgery. To obtain normal visual function, these patients needs surgery. Today, there are two different methods used for this condition; scleral suturing of the capsular complex or exchange of IOL to an iris-fixated IOL (Verisyse). In this study the investigators will look for advantages and dis-advantages for these two methods.

ELIGIBILITY:
Inclusion Criteria:

* patients with dislocation of IOL in the capsular complex who agree to participate in the study

Exclusion Criteria:

* patients with total dislocation of the capsular complex'
* patients with reduced general health
* patients who can't be randomized

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2020-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liv Drolsum, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Dalby M, Drolsum L, Kristianslund O. Repositioning surgery of different intraocular lens designs in eyes with late in-the-bag intraocular lens dislocation. J Cataract Refract Surg. 2021 Sep 1;47(9):1147-1152. doi: 10.1097/j.jcrs.0000000000000588. PMID 33754659
- [Derived] Kristianslund O, Ostern AE, Drolsum L. Astigmatism and Refractive Outcome After Late In-The-Bag Intraocular Lens Dislocation Surgery: A Randomized Clinical Trial. Invest Ophthalmol Vis Sci. 2017 Sep 1;58(11):4747-4753. doi: 10.1167/iovs.17-22723. PMID 28973318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Altogether 175 patients were assessed for eligibility, 104 patients were enrolled.
Groups:
- IOL Repositioning: Operation method: Intraocular lens repositioning by scleral suturing
  54 patients were randomised to this group. 11 patients were lost to follow-up before the 6-month postoperative visit because of serious illness and 1 death (unrelated to the condition studied).
- IOL Exchange: Operation method: Intraocular lens exchange with retropupillary iris-claw lens
  50 patients were randomised to this group. 8 patients were lost to follow-up before the 6-month postoperative visit because of serious illness (unrelated to the condition studied).
Period: Overall Study
Arm/Group | IOL Repositioning | IOL Exchange
Started | 54 | 50
Completed | 43 | 42
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IOL Repositioning | IOL Exchange | Total
Number analyzed (Participants) | 54 | 50 | 104
Age, Continuous [Mean (Full Range); unit: years] | 81 [56 to 94] | 82 [63 to 95] | 81.5 [56 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 63
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 50 | 104
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Norway | 54 | 50 | 104
Mean best-corrected visual acuity [Mean (Standard Deviation); unit: logMAR] | 0.37 (0.42) | 0.64 (0.77) | 0.50 (0.63)
Mean intraocular pressure [Mean (Standard Deviation); unit: mmHg] | 17.7 (5.0) | 18.3 (7.2) | 18.0 (6.2)
Mean time since cataract surgery [Mean (Standard Deviation); unit: years] | 10.6 (4.3) | 10.0 (4.3) | 10.3 (4.3)
Mean endothelial cell density [Mean (Standard Deviation); unit: cells/mm^2] | 1940 (418) | 1718 (449) | 1839 (444)

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity (BCVA)
Description: Measure for visual function. Measured in logMAR
Time Frame: 6 months, 1 year and 2 years
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | IOL Repositioning | IOL Exchange
Number analyzed (Participants) | 43 | 42
logMAR
  BCVA 6 months | 0.24 (0.29) | 0.35 (0.54)
  BCVA 1 year | 0.21 (0.26) | 0.23 (0.34)
  BCVA 2 years | 0.20 (0.29) | 0.22 (0.30)

2. Primary Outcome: Intraocular Pressure (IOP)
Description: Measure for the pressure inside the eye, measured with Goldman applanation tonometer, in mmHg.
Time Frame: 6 months and 2 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IOL Repositioning | IOL Exchange
Number analyzed (Participants) | 43 | 42
mmHg
  IOP 6 months | 16.5 (5.2) | 14.9 (4.2)
  IOP 2 years | 15.7 (4.0) | 14.1 (4.2)

3. Primary Outcome: Endothelial Density
Description: Corneal endothelial cell density (ECD), measured by confocal microscopy. Reported in cells per square millimeter
Time Frame: 6 months
Population: Some missing data due to inadequate corneal images
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | IOL Repositioning | IOL Exchange
Number analyzed (Participants) | 37 | 33
cells/mm^2 | 1858 (433) | 1514 (470)

4. Primary Outcome: Postoperative Complications
Description: Cystoid macular edema considered the most important long-term complication and therefore reported here.
Time Frame: 6 months and 2 years
Population: Some loss to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IOL Repositioning | IOL Exchange
Number analyzed (Participants) | 43 | 42
Participants
  CME 6 months: Cystoid macular edema | 3 | 4
  CME 6 months: No cystoid macular edema | 40 | 38
  CME 2 years: Cystoid macular edema | 5 | 6
  CME 2 years: No cystoid macular edema | 38 | 36

5. Secondary Outcome: Keratometry
Description: Keratometry of the cornea. Corneal astigmatism, measured in diopters.
Time Frame: 6 months (only analyzed/reported for this time frame)
Population: Some missing data due to poor image/measurement quality, overall number of participants therefore lower than the number of participants attending the 6-month visit
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | IOL Repositioning | IOL Exchange
Number analyzed (Participants) | 40 | 39
Diopters | 1.2 (1.0) | 1.2 (0.8)

6. Secondary Outcome: Questionnaire Visual Function-14 (VF-14) Score
Description: Questionnaire considering subjective visual function, scale 0-100 (higher scores mean better subjective visual outcome, lower scores means worse outcome).
Time Frame: 6 months (only analyzed/reported for this time frame)
Population: Some loss to follow-up
Measure: Mean (Standard Deviation); unit: score points
Arm/Group | IOL Repositioning | IOL Exchange
Number analyzed (Participants) | 43 | 42
score points | 91.6 (16.4) | 90.1 (18.2)

7. Secondary Outcome: IOL Location
Description: Measure IOL's location with slit lamp and Pentacam.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2020-12

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were registered as specific perioperative and postoperative complications related to the surgery.
  Otherwise we registered the number of participants that were lost to-follow up due to serious illness (other conditions than the studied) or death.
Arm/Group | IOL Repositioning | IOL Exchange
All-Cause Mortality (participants affected / at risk) | 1/54 | 0/50
Serious Adverse Events (participants affected / at risk) | 10/54 | 8/50
Other Adverse Events (participants affected / at risk) | 3/43 | 4/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IOL Repositioning (N=54) | IOL Exchange (N=50)
Serious illness (General disorders) | 10 (10) | 8 (8) — Serious adverse events were not related to intervention, "General disorders" were therefore chosen as a common term. The study population had a high age and therefore serious illness of some participants were anticipated
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IOL Repositioning (N=43) | IOL Exchange (N=42)
Cystoid macular edema (Eye disorders) | 3 (3) | 4 (4) — Postoperative complication, registered at the 6-month postoperative visit

LIMITATIONS AND CAVEATS:
Limitations to the study / the result:

Some loss to follow-up Some missing data for some of the parameters

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes